CLINICAL TRIAL: NCT00671385
Title: Early Screening of Breast Cancer Using Radiation-Free Pressure-Free Optical Scanning
Brief Title: Survey of Optical Values of the Breast Using Radiation-Free Pressure-Free Optical Scanning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spectros Corporation (Industry)
Collaborators: Stanford University (Other); University of California (Other); Palo Alto Medical Foundation (Other)
Responsible Party: Clinical Studies Manager, Spectros Corporation
Other Study IDs: BCA-003; CA126441; CA083597
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Breast Lesions; Breast Cyst; Early-Stage Breast Cancer; Benign Growth, Breast
Keywords: screening; compositional analysis; metabolism; breast; breast cyst; breast infection; breast inflammation; lipoma; benign growth; Women without a diagnosis for a region of interest in the breast
MeSH Terms: conditions — Breast Cyst; Breast Neoplasms; Mastitis; Lipoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women 21-50 years old: Women without a diagnosis of cancer or a history of cancer.

SUMMARY:
The purposes of this study is to establish normal optical values of breast tissue in the general population. This will allow for establishing normals for breast composition, and is expected to be useful in the classification of breast lesions into groups such as cysts, benign growths, inflammatory lesions, and possibly early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* You must be female
* You must be 21 to 50 years old
* You must not have or have had breast cancer.
* You must not have or have had breast implants or breast surgery
* You must not have had a breast biopsy or injury, or a breast infection, in 90 days.

Exclusion Criteria:

* Any one or more of the above conditions not met
* Lack of informed consent

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 18-50 with who EITHER (a) have a region of interest but without a diagnosis, or (b) are healthy volunteers without breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Optical normals for the breast for a variety of conditions | 3 years

SECONDARY OUTCOMES:
Diagnostic compositional standards for (a) diagnosis of a condition such as cyst, benign growth, inflammation, and/or (b) referral for additional evaluation of a region of interest. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David A Benaron, MD, Study Director — Spectros Corporation
Locations (1):
- Spectros Corporation, Portola Valley, California, United States